CLINICAL TRIAL: NCT03361449
Title: Effect of Flamingo Exercises on Balance in Patients With Balance Impairment Due to Senile Osteoarthritis
Brief Title: Effect of Flamingo Exercises on Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, ASLIHAN UZUNKULAOGLU, Ufuk University Faculty of Medicine Ethical Comitee, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30112015-7
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis; Gait Disorders, Neurologic
MeSH Terms: conditions — Osteoarthritis; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): training with kinesthetic ability trainer.
  Interventions: Other: training with kinesthetic ability trainer
- Group 2 (Active Comparator): Flamingo exercise
  Interventions: Other: Flamingo exercise
- Group 3 (Active Comparator): training with kinesthetic ability trainer and Flamingo exercise
  Interventions: Other: Flamingo exercise; Other: training with kinesthetic ability trainer

INTERVENTIONS:
Other: Flamingo exercise — Flamingo exercise
  Arms: Group 2; Group 3
Other: training with kinesthetic ability trainer — training with kinesthetic ability trainer
  Arms: Group 1; Group 3

SUMMARY:
The aim of this study is to determine the effect of flamingo exercise on balance in patients with balance impairment due to senil osteoarthritis

DETAILED DESCRIPTION:
Changes in the sensory, neurological, and musculoskeletal systems in older adults affect several motor tasks,including postural balance. Also osteoarthritis contribute to this process. Older people can gain balance disorders. The flamingo balance exercise is a full lower body workout utilizing many major muscle groups. Therefore investigators aimed to determine the effect of flamingo exercise combined with kinesthetic ability trainer or alone in patients with balance impairment due to osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years old
* osteoarthritis diagnosis
* Balance impairment (Berg balance scale 21-40 points)

Exclusion Criteria:

* Severe neurological deficit
* Defect of vision
* Vitamin B12 deficiency
* Sedative drug use

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-25 (Estimated); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
kinesthetic ability trainer static score | 4 weeks
  kinesthetic ability trainer static score
kinesthetic ability trainer static dynamic score | 4 weeks
  kinesthetic ability trainer static dynamic score
Berg Balance Scale | 4 weeks
  a scale for balance
Timed up and Go test | 4 weeks
  for balance and gait
activity specific balance scale. | 4 weeks
  for balance

IPD SHARING:
Plan to Share IPD: No